CLINICAL TRIAL: NCT01857557
Title: Evaluation of an Aerobic Exercise Program in Migraine Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges with participant recruitment as a result of COVID-19 pandemic
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Farnaz Amoozegar, Dr Farnaz Amoozegar, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24702
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Migraine
Keywords: Exercise; Fitness program
MeSH Terms: conditions — Migraine Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise (Experimental): Fitness program for migraine patients in addition to usual headache care.
  Interventions: Other: Aerobic exercise
- Control Group (No Intervention): Patients receiving usual headache care but no exercise program

INTERVENTIONS:
Other: Aerobic exercise — Patients receiving exercise program in addition to usual headache care
  Arms: Aerobic Exercise

SUMMARY:
This trial assesses the impact of a supervised aerobic exercise program by a kinesiologist in patients with migraine. Patients can be assigned to one of two groups 1)The exercise group or 2)non-exercise group. This is a important area to study because there is currently limited information regarding exercise and its impact on migraine frequency and severity. In many cases, migraine patients are disabled by their headaches and sometimes will not have a significant response to medications. As a result, it is important to study other non-pharmacological interventions. In this study, the investigators hope to show the benefits of exercise by a reduction in number of headache days per month as well as by improvement in quality of life, disability,depression,anxiety,and aerobic fitness.This study will not interfere with the usual treatment patients receive at our headache clinic and patients can remain on medications deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet diagnostic criteria for migraine without aura, migraine with aura or chronic migraine.
2. Patients must be 18-50 years of age.
3. Individuals motivated to exercise and complete the study.

   -

Exclusion Criteria:

1. Patient has a headache on more than 25 days a month
2. Patient is a medication over-user by International Headache Society (IHS) criteria
3. Patient currently has a fitness program with regular aerobic exercise for 30 minutes three times a week or more.
4. Known cardiovascular disease which contraindicates the exercise program
5. Inability to complete the outcome measure questionnaires. -

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-08; Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Days with headache per month (based on headache diaries),comparing the change from baseline to month 3 and 6 post-randomization in the control versus the intervention group. Migraine Specific Quality of Life Questionnaire scores | At baseline,3, 6 months

SECONDARY OUTCOMES:
Show Improvement in measures of quality of life,disability,depression,anxiety,and aerobic fitness | Baseline, 3 ,6 months post randomization
  Headache Impact Test (HIT-6 )score, Migraine Disability Assessment scores, Patient Health Questionnaire(PHQ-9 )scores,Generalized Anxiety Disorder (GAD-7) scores, Average headache intensity, Body Mass Index, Aerobic fitness

OTHER OUTCOMES:
Adherence to fitness program in the intervention group | At 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Dr Farnaz Amoozegar, MD, FRCPC, Principal Investigator — South Health Campus, Calgary, Alberta, Canada
Locations (1):
- South Health Campus, Calgary, Alberta, Canada